CLINICAL TRIAL: NCT05176158
Title: Efficacy of Dexketoprofen Prescribed According to the Circadian Rhythms
Brief Title: Dexketoprofen Dosage According to Chronotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-000736-26
Record Dates: First submitted 2021-12-14; First posted 2022-01-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2022-10

CONDITIONS: Tooth, Impacted; Trismus; Pain; Inflammatory Response
Keywords: Third; Dexketroprofen; Randomized
MeSH Terms: conditions — Tooth, Impacted; Trismus; Pain | interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning dosage (Experimental): Dexketoprofen pill at morning; Placebo at night
  Interventions: Drug: Dexketoprofen 25 MG
- Night dosage (Experimental): Placebo pill at morning; Dexketoprofen at night
  Interventions: Drug: Dexketoprofen 25 MG

INTERVENTIONS:
Drug: Dexketoprofen 25 MG — Pill at morning
  Other Names: Morning dosage
  Arms: Morning dosage
Drug: Dexketoprofen 25 MG — Pill at night
  Other Names: Night dosage
  Arms: Night dosage

SUMMARY:
Lower third molar extraction is one of the most common treatments in oral surgery practice. It is a treatment with inherent complications such as postoperative pain, swelling or trismus. In order to minimize disconfort after extraction, analgesic and anti-inflammatory medication is prescribed. Recently, it is seen that circadian rhythm may play an important role on drugs metabolism, modulating its effect depending on the moment of administration.

The aim of the study is to analyze if dosage modification of a Non Steroideal Anti-Inflammatory (dexketoprofen) affects on postoperative pain, swelling and open mouth limitation according the circadian clock

DETAILED DESCRIPTION:
A randomized crossover split-mouth clinical trial will be performed. After third molar extractions, patients will be prescribed randomly in one side intake morning medication dosage while the contralateral side will be prescribed a night dosage. Moreover, a blood sample will be obtained to analyze the inflammatory profile.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral impacted lower third molar

Exclusion Criteria:

* NSAID allergic
* Contraindication of surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Post operatory pain | From the day of the surgical procedure to the seventh-day
  Postoperatory pain with Visual Analogue Scale (VAS: 0 (no pain) to 10 (worst pain))

SECONDARY OUTCOMES:
Swelling | Baseline and post operatory (day 1, day 3, day 7)
  Distance from tragus to pogonion

OTHER OUTCOMES:
Trismus | Baseline and post operatory (day 1, day 3 and day 7)
  Open mouth limitation in milimiters, interincisal distance
Inflammatory profile for IL-1B, IL-6, IL-8, IL-10, TNF alpha | Baseline, day 3 and day 7
  Blood sample analysis for inflammatory cytokines in IU/ml by ELISA test (enzyme-linked immunoassay)

CONTACTS AND LOCATIONS:
Locations (1):
- UCM, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Gonzalez F, Abusamak M, Ruiz LV, Saez-Alcaide LM, Al-Waeli H, Tamimi F, Garcia-Denche JT. Dexketoprofen Time-Dependent Administration After Third Molar Extraction: A Pilot Randomized Cross-Over Controlled Trial. Clin Exp Dent Res. 2026 Feb;12(1):e70163. doi: 10.1002/cre2.70163. PMID 41510697